CLINICAL TRIAL: NCT04974970
Title: Pilot Study on Immunotherapy for the Treatment of Persistant Peanut Allergy
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: early termination due to insufficient recruitment
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Jean-Christoph Caubet, Principal investigator, University Hospital, Geneva
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018-02316
Record Dates: First submitted 2021-07-16; First posted 2021-07-23 (Actual); Last update posted 2023-08-28 (Actual); Status verified 2023-08

CONDITIONS: Food Allergy; Peanut Allergy
MeSH Terms: conditions — Food Hypersensitivity; Peanut Hypersensitivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Peanut allergenic extract (Experimental): injected peanut extract.
  Interventions: Drug: Peanut Immunotherapy

INTERVENTIONS:
Drug: Peanut Immunotherapy — Treatment will be injected peanut extract every 2 weeks for a period of 3 months.

SUMMARY:
The purpose of this trial is to assess the safety and efficacy of peanut immunotherapy in children and adults with peanut allergy. Participants will receive immunotherapy with peanut every 2 weeks for a period of 3 months.

ELIGIBILITY:
Inclusion Criteria:

1. Informed Consent as documented by signature.
2. Male or female subjects 12 to 45 years old at screening visit.
3. Patients with convincing history of IgE-mediated systemic allergic reaction after consumption of peanut, and specific IgE above 95% positive predictive value:

   a. Peanut ≥ 15kU/L or Ara h 2 ≥ 5U/L
4. Patients without a convincing history of IgE-mediated systemic allergic reaction (for example only oral symptoms) after consumption of peanuts but with clear evidence of sensitization (SPT > 3 mm and/or positive specific IgE (> 0.1kU/l) and a positive standardized food challenge to peanut between V0 and V1.

Exclusion Criteria:

1. Subjects with a history of severe anaphylaxis to the incriminated food with the following symptoms: hypotension, hypoxia, neurological compromise (collapse, loss of consciousness or incontinence).
2. Subjects with a history of systemic reaction to peanutskin prick test with commercial extract.
3. Uncontrolled asthma (Forced expiratory volume at one second (FEV1) <70% of predicted value), active eosinophilic oesophagitis or any condition deemed incompatible by the investigator.
4. Known or suspected systemic mastocytosis.
5. Subject currently under allergen immunotherapy.
6. Subject/parent with excessive anxiety unlikely to cope with study conditions as per investigator's opinion.
7. Participation in a clinical study with a new investigational drug within the last 3 months or for a biological within the last 6 months prior to or during the study.
8. Use of immunosuppression or immunomodulatory drug (including anti-IgE or anti-Tumor necrosis factor (TNF)) within 1 year prior to inclusion in study.
9. Relative counter-indication or inability to use epinephrine auto-injector.
10. Subjects receiving beta-blockers or angiotensin converting-enzyme (ACE) inhibitors.
11. Women who are pregnant or breast feeding.
12. Intention to become pregnant during the course of the study, or inadequate contraceptive measures for women of child-bearing age (contraceptive measures considered adequate are: intrauterine devices, hormonal contraceptives, such as contraceptive pills, implants, transdermal patches, hormonal vaginal devices or injections with prolonged release).
13. Other clinically significant concomitant disease states (e.g., renal failure, hepatic dysfunction, cardiovascular disease, etc.).
14. Diseases with a contraindication for the use of adrenalin (e.g. hyperthyroidism, glaucoma).
15. Known or suspected non-compliance, drug or alcohol abuse.
16. Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia, etc. of the participant.
17. Patients who are employees of the sponsor, institution or 1st grade relatives or partners of the investigators

Ages: 12 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 12 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2022-04-19 (Actual); Study Completion 2022-04-19 (Actual)

PRIMARY OUTCOMES:
Result (positive or negative) and cumulative reaction threshold at 3 months peanut oral food challenge (OFC). | 3 months
  An unblinded evaluation of peanut OFC cumulative reaction threshold after 3 months of peanut immunotherapy.

SECONDARY OUTCOMES:
Change in serum levels of allergen specific IgE and IgG4 after 6 weeks and 3 months of treatment compared to baseline peanut specific IgE and IgG4 after 3 months of treatment with peanut extract. | 3 months
  An evaluation of changes in serum levels of allergen specific IgE and IgG4 after 6 weeks and 3 months of treatment compared to baseline peanut specific IgE and IgG4 after 3 months of treatment with peanut extract.
Change in titrated skin prick test after 6 weeks and 3 months of treatment with peanut extract compared to baseline. | 3 months
  An evaluation of changes in titrated skin prick tests after 6 weeks and 3 months of treatment with peanut extract compared to baseline.
Incidence rate of treatment emergent adverse events during peanut immunotherapy | 3 months
  An unblinded evaluation of the safety of peanut immunotherapy as measured by the incidence of treatment-emergent adverse events (AEs and SAEs).

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Christoph Caubet, MD, Principal Investigator — University Hospitals of Geneva
Locations (1):
- Pediatric allergy unit, Hôpitaux Universitaires de Genève (HUG), Geneva, Switzerland